CLINICAL TRIAL: NCT05873218
Title: Impact of Prophylactic Ephedrine on Fetal Heart Tracing and Uterine Tetanic Contraction After Combined Spinal Epidural on Laboring Parturients
Brief Title: Impact of Prophylactic Ephedrine on Fetal Heart Tracing and Uterine Tetanic Contraction After CSE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Vice Chair of Education Department of Anesthesiology, Pain, & Perioperative Medicine Icahn School of Medicine at Mount Sinai Director of Education Mount Sinai HELPS Center, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY-22-01334
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Labor
Keywords: Randomized Control Trial; Prophylactic Ephedrine; Fetal Heart Rate Tracing; Combined Spinal Epidural; Labor analgesia
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ephedrine (Experimental): 3 minutes after the placement of a combined spinal epidural with 25 mcg fentanyl, 7.5 mg ephedrine IV will be administered to the patient, 12 minutes later, a second dose of 7.5mg will be administered to the patient as long as the patient is not hypertensive (BP no greater than 140/90)
  Interventions: Drug: Ephedrine
- Placebo (Placebo Comparator): 3 minutes after the placement of a combined spinal epidural with 25 mcg fentanyl, 2.5cc 0.9% NS IV will be administered to the patient, 12 minutes later, a second dose of , 2.5cc 0.9% NS will be administered to the patient.
  Interventions: Drug: Normal Saline Placebo

INTERVENTIONS:
Drug: Ephedrine — The intervention will be up to two 7.5 mg doses of ephedrine given after the placement of a combined spinal epidural with 25 mcg intrathecal fentanyl timed 3 and 15 minutes after intrathecal opiate administration.
  Arms: Ephedrine
Drug: Normal Saline Placebo — Placebo will be administered at matching rate.
  Arms: Placebo

SUMMARY:
Labor analgesia is an important component of the care of laboring patients. A known side effect of combined spinal and epidural anesthesia (a type of labor analgesia) is an increased incidence of category II fetal heart rate tracing (defined below) and low blood pressure. The study team aims to study if a prophylactic dose of ephedrine will decrease the occurrence of this type of tracing after combined spinal epidural (CSE) anesthesia placement. Ephedrine is not currently routinely used as prevention for category II tracings or low blood pressure. The use of Ephedrine in this study is investigational (this is the first time that the drug has been studied for its effect on these conditions).

Fetal heart rate (FHR) tracings are classified into three categories. In clinical practice, FHR tracing categories are used as a guide to obstetric management and suggest the following approach:

* Category I tracing is "reactive" and reassuring → may continue labor
* Category II tracing is neither category I nor category III. For obvious reasons, category II is the broadest and largest category, consisting of various FHR tracing patterns that do not fit into either category I or category III.
* Category III tracing is non-reassuring → expedited vaginal or cesarean delivery recommended.

A Category II tracing is not diagnostic. Most pregnancies have at least one Category II tracing. There is not always an identifiable reason for a Category II tracing.

Ephedrine is a medication that causes an increase in heart rate and blood pressure while also causing some degree of relaxation of the uterus therefore improving uterine blood flow. It has been used in the obstetric population for over 50 years without issues. The dose that the research team will administer, 7.5 mg, is below the dose the research team will often administer to treat hypotension (low blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-55 years
* Requesting labor analgesia
* Able to provide informed written consent
* Category 1 fetal tracing prior to placement of neuraxial anesthesia

Exclusion Criteria:

* Refusal of neuraxial anesthesia
* History of hypertension
* Suspected pre-eclampsia
* Category 2 or 3 fetal tracing prior to placement of neuraxial anesthesia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of category II fetal heart rate tracing | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of category II fetal heart rate tracing up to 30 minutes after administration of intrathecal opiate

SECONDARY OUTCOMES:
Incidence of uterine tetanic contractions | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of uterine tetanic contractions after combined spinal epidural placement
Incidence of uterine hypertorus | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of uterine hypertorus up to 30 minutes after administration of intrathecal opiate
Incidence of fetal bradycardia | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of fetal bradycardia up to 30 minutes after administration of intrathecal opiate
Incidence of rescue administration of ephedrine, terbutaline, or nitroglycerin | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of rescue administration of ephedrine, terbutaline, or nitroglycerin up to 30 minutes after administration of intrathecal opiate
Incidence of antihypertensive treatment after ephedrine administration | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of antihypertensive treatment after ephedrine administration
Incidence of urgent/emergent cesarean delivery | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of urgent/emergent cesarean delivery within 30 minutes of intrathecal opiate administration
Incidence of hypotension | day 1, 30 minutes after administration of intrathecal opiate
  Incidence of hypotension as defined as systolic blood pressure decrease of 20% versus baseline, systolic blood pressure under 90 mmHG, or symptoms of hypotension such as light headedness
Average HR changes | day 1, 30 minutes after administration of intrathecal opiate
  Average HR changes 30 minutes after intrathecal opiate administration
Average blood pressure changes | day 1, 30 minutes after administration of intrathecal opiate
  Average blood pressure changes 30 minutes after intrathecal opiate administration of systolic and diastolic blood pressure
Number of patients with systolic blood pressure under 90 mmHG | End of study, at 6 months
  Systolic blood pressure under 90 mmHG, or symptoms of hypotension such as light headedness

CONTACTS AND LOCATIONS:
Overall Officials: James Leader, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount SInai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be protected.